CLINICAL TRIAL: NCT03403595
Title: Safety and Dosimetry of 177Lu-EB-PSMA617 in Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: 177Lu-EB-PSMA617 in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH-NM16; ZIAEB000073 (NIH)
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — 177Lu-EB-PSMA-617

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-EB-PSMA-617 dosimetry calculation (Experimental): All patients were intravenous injected with single dose 0.80-1.1 GBq (21.5-30 mCi) of 177Lu-EB-PSMA-617, then monitored at 2, 24, 72, 120 and 168 hours post-injection.
  Interventions: Drug: 177Lu-EB-PSMA-617

INTERVENTIONS:
Drug: 177Lu-EB-PSMA-617 — accepted intravenous injection of 177Lu-EB-PSMA-617 and monitored at 2, 24, 72, 120 and 168 hours post-injection.

SUMMARY:
This is an open-label, non-controlled, non-randomized study to assess the safety and measure image-based absorbed dose of 177Lu-EB-PSMA-617 in patients with metastatic castration-resistant prostate cancer (mCRPC) who will undergo radioliagnd therapy using 177Lu-EB-PSMA-617. All patients underwent whole-body 68Ga-PSMA PET/CT for selection and accepted intravenous injection with single dose 0.80-1.1 GBq (21.5-30 mCi) of 177Lu-EB-PSMA-617 within one week, then monitored at 2, 24, 72, 120 and 168 h after 177Lu-EB-PSMA617 administration with serial whole body planar and SPECT/CT imaging.

DETAILED DESCRIPTION:
Prostate cancer is the most frequent malignant tumor in men worldwide. Prostate-specific membrane antigen (PSMA), is a surface molecule specifically expressed by prostate tumors which was shown to be a valid target for radiotherapy. 177Lu-PSMA-617, a urea-based compound, provide an effective target for the treatment of metastatic castration-resistant prostate cancer. However, a major problem in the therapeutic use of 177Lu-PSMA-617 has been its short half-life and fast rate of clearance. This study was designed to investigate the safety, dosimetry and preliminary effects of 177Lu-EB-PSMA-617 in patients with metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* All the patients had progressive metastatic castration-resistant prostate cancer that did not respond to androgen-suppression therapy and/or systemic chemotherapy. Distant metastases with high PSMA expression were confirmed on 68Ga-PSMA PET/CT within one week before the injection of 177Lu-EB-PSMA-617.

Exclusion Criteria:

* The exclusion criteria were a serum creatinine level of more than 150 μmol per liter, a hemoglobin level of less than 10.0 g/dl, a white-cell count of less than 4.0× 109/L, a platelet count of less than 100 × 109/L, a total bilirubin level of more than 3 times the upper limit of the normal range and a serum albumin level of more than 3.0 g per deciliter, cardiac insufficiency including carcinoid heart valve disease, a severe allergy or hypersensitivity to radiographic contrast material, claustrophobia, and pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 177Lu-EB-PSMA617 in normal organs and metastatic castration-resistant prostate cancer. | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value at each time point in normal organs and metastatic castration-resistant prostate cancer will be measured

SECONDARY OUTCOMES:
Adverse events collection | 2 months
  Adverse events within 2 months after the injection and scanning of patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD,PHD, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China